CLINICAL TRIAL: NCT00718939
Title: Rheos® Diastolic Heart Failure Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 360014
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Diastolic Heart Failure
Keywords: Diastolic Heart Failure; Cardiac dysfunction; Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rheos ON (Other): Study participants in this arm will have the device turn on for six months and remains on.
  Interventions: Device: Rheos Baroreflex Activation Therapy System
- Rheos OFF (Other): Study participants in this arm will have the device turned off for 6 months and then turned on.
  Interventions: Device: Rheos Baroreflex Activation Therapy System

INTERVENTIONS:
Device: Rheos Baroreflex Activation Therapy System — The two (2) Rheos Carotid Sinus Leads conduct the activation energy from the Rheos Implantable Pulse Generator to the baroreceptors located on the left (Left Carotid Sinus Lead) and right (Right Carotid Sinus Lead) carotid sinus. This energy activates the baroreflex by inducing signals that the brain interprets as elevated blood pressure.

SUMMARY:
The CVRx® Rheos® Diastolic Heart Failure Trial is a prospective, randomized, double blind trial with up to 60 subjects conducted at up to five centers in Europe. All subjects will be followed up to one year post implant.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age.
* Have bilateral carotid bifurcations that are below the level of the mandible.
* Have a left ventricular ejection fraction ≥ 45%.
* Clinical Heart Failure with elevated BNP or NT-Pro-BNP.

Exclusion Criteria:

* History of or suspected baroreflex failure or autonomic neuropathy.
* History of symptomatic bradyarrhythmias, pericardial constriction, infiltrative cardiomyopathy, cardiac valvular disease.
* Organ or hematologic transplant.
* History of prior surgery, radiation, or stent placement in carotid sinus region.
* History of severe chronic kidney disease.
* Life expectancy to less than one year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Assess left ventricular mass index (LVMI). | at six months post- randomization.
Assess safety by evaluating all adverse events. | through six months post -implant

SECONDARY OUTCOMES:
To assess difference between randomization groups in blood pressure changes, blood levels and quality of life. | six months post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian A Pichlmaier, MD, Principal Investigator — Medizinische Hoschschule Hannover; Johannes Sperzel, MD, Principal Investigator — Kerckhoff-Klinik Forschungsgesellschaft mbH; Prof. Uta Hoppe, MD, Principal Investigator — University of Cologne; Herbert Naegele, MD, Principal Investigator — Krankenhaus Reinbek St.Adolfsstif
Locations (4):
- Germany (4):
  - Kerckhoff-Klinik Forschungsgesellschaft mbH, Bad Nauheim
  - University of Cologne, Cologne
  - Krankenhaus Reinbek St.Adolfsstif, Hamburg-Reinbek
  - Medizinische Hoschschule Hannover, Hanover

REFERENCES:
- See also: Related Info — http://www.cvrx.com